CLINICAL TRIAL: NCT02006901
Title: Comparative Effectiveness of Microdecompression and Laminectomy for Central Lumbar Spinal Stenosis - An Observational Study
Brief Title: Comparative Effectiveness of Microdecompression and Laminectomy for Central Lumbar Spinal Stenosis
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/643
Record Dates: First submitted 2013-12-02; First posted 2013-12-10 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Spinal Stenosis; Spinal Cord Compression
Keywords: surgical procedures, operative; lumbar vertebrae; decompression, surgical; microdecompression; laminectomy; registries
MeSH Terms: conditions — Spinal Stenosis; Spinal Cord Compression | interventions — Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- microdecompression: surgical microdecompression using a bilateral or unilateral approach depending on the surgeon's preference and the individual patient's anatomy and symptoms.
  Interventions: Procedure: microdecompression
- laminectomy: the spinous process and the laminae of the involved level(s) as well as the medial aspects of the facet joints are resected
  Interventions: Procedure: laminectomy

INTERVENTIONS:
Procedure: microdecompression — a minimal invasive surgical technique
  Groups: microdecompression
Procedure: laminectomy — The traditional open surgical technique: decompression with removal of the spinous process, lamina and often the medial facets
  Groups: laminectomy

SUMMARY:
Introduction: This observational study is designed to test the equivalence between the clinical effectiveness of microdecompression and laminectomy in the surgical treatment of central lumbar spinal stenosis. Lumbar spinal stenosis is the most frequent indication for spinal surgery in the elderly, and as the oldest segment of the population continues to grow its prevalence is likely to increase. However, data on surgical outcomes are limited. Open or wide decompressive laminectomy, often combined with medial facetectomy and foraminotomy, was formerly the standard treatment. In recent years a growing tendency towards less invasive decompressive procedures has emerged. Many spine surgeons today perform microdecompression for central lumbar spinal stenosis.

Prospectively registered treatment and outcome data are obtained from the Norwegian Registry for Spine Surgery (NORspine).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of central lumbar spinal stenosis
* Operation in ≤2 lumbar levels with either open decompressive laminectomy, bilateral microdecompression or unilateral microdecompression for bilateral decompression in the time period between October 2006 and December 2011
* Included in the NORspine registry

Exclusion Criteria:

* History of lumbar fusion
* Previous surgery in the lumbar spine
* Discectomy as part of the decompression
* Associated pathological entities such as disc herniation, spondylolisthesis or scoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had operation in ≤2 lumbar levels with either open decompressive laminectomy, bilateral microdecompression or unilateral microdecompression for bilateral decompression in Norway in the time period between October 2006 and December 2011
Sampling Method: Non-Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
change in Oswestry Disability Index | between baseline and 12-months follow-up
  collected through the Norwegian Registry for Spine Surgery (NORspine)

SECONDARY OUTCOMES:
changes in health-related quality of life | between baseline and 12-months follow-up
  measured by Euro-Qol-5D, collected through the Norwegian Registry for Spine Surgery (NORspine)
patient reported post-operative complications | 3 months
  wound infection, urinary tract infection, pneumonia, pulmonary embolism, and deep venous thrombosis
surgeon reported complication | reported at discharge (expected average hospital stay of 3 days)
  intraoperative hemorrhage requiring blood replacement, unintentional durotomy, cardiovascular complications, respiratory complications, anaphylactic reactions, and wrong level surgery
Length of hospital stay | reported at discharge (expected average hospital stay of 3 days)
  Length of hospital stay before discharge
Length of surgery | reported at discharge (expected average hospital stay of 3 days)
  Length of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Gulati, MD, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Nerland US, Jakola AS, Solheim O, Weber C, Rao V, Lonne G, Solberg TK, Salvesen O, Carlsen SM, Nygaard OP, Gulati S. Minimally invasive decompression versus open laminectomy for central stenosis of the lumbar spine: pragmatic comparative effectiveness study. BMJ. 2015 Apr 1;350:h1603. doi: 10.1136/bmj.h1603. PMID 25833966
- [Derived] Nerland US, Jakola AS, Solheim O, Weber C, Rao V, Lonne G, Solberg TK, Salvesen O, Carlsen SM, Nygaard OP, Gulati S. Comparative effectiveness of microdecompression and laminectomy for central lumbar spinal stenosis: study protocol for an observational study. BMJ Open. 2014 Mar 20;4(3):e004651. doi: 10.1136/bmjopen-2013-004651. PMID 24650809